CLINICAL TRIAL: NCT03875560
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Safety, Pharmacokinetic, Pharmacodynamic and Preliminary Efficacy Study of IC14 in Adult Patients With Dengue Fever
Brief Title: IC14 in Adult Patients With Dengue Fever
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: seeking funding
Sponsor: Implicit Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: EDF-01
Record Dates: First submitted 2016-08-16; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A/Single Dose (Experimental): IC14 0.5, 1.0 or 2.0 mg/kg IV as a single dose (subjects are assigned and not randomized to this arm. When Part A is complete, Enrollment to Part B will commence).
  Interventions: Biological: IC14
- Part B/Cohort 1 (Experimental): IC14 4 mg/kg/day IV or placebo IV x 1 day.
  Interventions: Biological: IC14; Drug: Placebo
- Part B/Cohort 2 (Experimental): IC14 8 mg/kg/day IV or placebo IV x 1 day.
  Interventions: Biological: IC14; Drug: Placebo
- Part B/Cohort 3 (Experimental): IC14 2 mg/kg/day IV x 1 day followed by IC14 1 mg/kg/day IV x 3 days or placebo IV daily for 4 days.
  Interventions: Biological: IC14; Drug: Placebo
- Part B/Cohort 4 (Experimental): IC14 4 mg/kg/day IV x 1 day followed by IC14 2 mg/kg/day IV x 3 days or placebo IV daily for 4 days.
  Interventions: Biological: IC14; Drug: Placebo

INTERVENTIONS:
Biological: IC14 — recombinant chimeric anti-human CD14 monoclonal antibody
Drug: Placebo — Inactive
  Arms: Part B/Cohort 1; Part B/Cohort 2; Part B/Cohort 3; Part B/Cohort 4

SUMMARY:
Randomized, double-blind, placebo-controlled, safety, PK/PD and preliminary efficacy study of intravenous IC14 in adult patients in a dengue-endemic region presenting with fever > 38°C for < 48 hours with a positive NS1 strip assay or reverse-transcriptase polymerase chain reaction assay for dengue virus.

DETAILED DESCRIPTION:
The study will be conducted in two parts and will include an open label phase of a single dose of IC14 (Part A) and a randomized phase of multiple doses of IC14 and placebo (Part B). Up to 52 patients will be enrolled in both parts of the study.

Part A will consist of 12 patients given one of three doses of IC14 as a single dose open-label . Each patient must complete 14 days before the enrollment of subsequent patients. Part A subjects will be hospitalized for 4 days. During and at the end of 4-day admission to the clinical research unit, and on Study Days 5, 6, 7, 14, 21 and 32, Part A patients will have their health status assessed. The last subject in Part A must complete 32 days of participation before Part B of the trial is opened.

Part B consists of 40 patients randomized equally to one of 4 dosing regimens which will include a single dose or multiple doses of IC14 or placebo given at different dosing frequencies. In Part B, Cohort 1 and 2 subjects (single dose) will be inpatient for 4 days and Cohort 3 and 4 subjects (four daily doses) will be inpatient for 5 days. During and at the end of the admission to the clinical research unit, and on Study Days 5, 6, 7, 14, 21 and 32, Part B patients will have their health status assessed.

ELIGIBILITY:
Inclusion Criteria

* Fever > 38°C for < 48 hours and clinical presentation consistent with dengue fever.
* Positive NS1 strip assay or reverse-transcriptase polymerase chain reaction (RT-PCR) assay for dengue virus.
* Informed consent form signed and dated by the patient.
* Subject able to give informed consent and able to comply with all study visits and all study procedures.
* Females of childbearing potential should be using and committed to continue using acceptable birth control methods.

  * Sexual abstinence (inactivity) for 1 month prior to screening through study completion; or
  * Intrauterine device (IUD) in place for at least 3 months prior to study through study completion; or
  * Stable hormonal contraception for at least 3 months prior to study through study completion; or
  * Surgical sterilization (vasectomy) of male partner at least 6 months prior to study.
* To be considered of non-childbearing potential, females should be surgically sterilized (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 2 months prior to study) or be post-menopausal and at least 3 years since last menses.

Exclusion Criteria

* One or more of the following dengue warning signs and symptoms:

  * Intense and continuous abdominal pain (referred pain or on palpation);
  * Persistent vomiting;
  * Fluid accumulation (ascites, pleural effusion, or pericardial effusion);
  * Postural hypotension and/or collapse;
  * Painful hepatomegaly > two centimeters below the right costal margin;
  * Mucosal bleeding;
  * Major bleeding (hematemesis and/or melena);
  * Lethargy and/or irritability;
  * Diminished urine output;
  * Hypothermia;
  * Progressive increase in hematocrit or 20% above baseline or normal for age;
  * Abrupt drop in platelets;
  * Respiratory discomfort.
* One or more of the following signs and symptoms of severe dengue, such as:

  * Severe plasma extravasation, leading to shock evidenced by one or more of the following:
  * Tachycardia;
  * Cold distal extremities;
  * Weak, thready pulse;
  * Slow capillary refill (> 2 seconds);
  * Pulse pressure < 20 mmHg;
  * Tachypnea; or
  * Oliguria (<1.5 mL/kg/hr).
  * Systolic blood pressure < 90 mmHg or decrease >40 mmHg;
  * Cyanosis;
  * Fluid accumulation with respiratory discomfort;
  * Severe bleeding; or
  * Severe organ impairment, evidenced by one or more of the following:
  * Liver impairment (AST >1000 U/L, international normalized ratio >1.5);
  * Renal impairment (serum creatinine ≥1.5 mg/dL); or
  * Myocarditis, pericarditis, or clinical heart failure (by chest x-ray, echocardiography, electrocardiogram, or cardiac enzymes if available).
* Female who is pregnant, lactating or of childbearing potential.
* Self-reported or suspected congenital or acquired immunodeficiency (including HIV infection); or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the previous 3 months).
* Prior vaccination against dengue fever.
* Significant chronic illness that, in the opinion of the Investigator, would interfere with study validity, conduct or completion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety, tolerability) | 32 days
  Number of patients with treatment-related adverse events as classified according to MedDRA
Area under the curve of IC14 serum concentration | 14 days
  Area under the curve of IC14 serum concentration

SECONDARY OUTCOMES:
Dengue viral load | 32 days
  Impact of treatment on dengue viral load measured by quantitative viral load and plasma NS1 viral protein
Fever | 32 days
  Impact of treatment on duration of fever
Dengue symptom score | 32 days
  Impact of treatment on dengue symptom severity (0 normal] to 24 [worst])
Disease severity | 32 days
  Impact of treatment on duration of hospitalization; incidence and duration of intensive care unit admission; and incidence of progression to dengue with warning signs or severe dengue
Mortality | 32 days
  Impact of treatment on survival

CONTACTS AND LOCATIONS:
Overall Officials: Jan Agosti, MD, Study Director — Implicit Bioscience

IPD SHARING:
Plan to Share IPD: Undecided